CLINICAL TRIAL: NCT04631393
Title: Patient-controlled Sedation in Port Implantation (PACSPI-1)-a Feasibility Trial
Brief Title: Patient-controlled Sedation in Port Implantation (PACSPI-1)
Acronym: PACSPI-1
Status: Completed | Type: Observational
Sponsor: Stefanie Seifert (Other Government)
Responsible Party: Sponsor-Investigator, Stefanie Seifert, Principal Investigator, Region Jönköping County
Organization: Region Jönköping County (Other Government)
Other Study IDs: EPM 2020-02642
Record Dates: First submitted 2020-11-10; First posted 2020-11-17 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Pain; Patient Satisfaction
Keywords: patient-controlled sedation; totally implantable venous access devices; subcutaneous implanted venous port; local anesthesia; propofol; alfentanil; indwelling catheter
MeSH Terms: conditions — Pain; Patient Satisfaction | interventions — Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Propofol Alfentanil — Propofol and Alfentanil are self-administered by the participant.
  Other Names: Propofol/Alfentanil self-administration

SUMMARY:
The purpose of this prospective, observational study is to assess the feasibility of patient-controlled sedation (PCS) for implantation of subcutaneous venous ports (SVP).

DETAILED DESCRIPTION:
The main objective of this trial is to study the feasibility of (PCS) with propofol and alfentanil during SVP implantation.

Participants included in the study are able to administer a combination of propofol and alfentanil using a patient-controlled sedation pump. This allows the patient to self-control their sedation/analgesia during SVP implantation. The pump enables the patient via a hand-held button to trigger the release of a single bolus. A bolus of 0.5ml programmed into the pump contains a combination of 4.5mg propofol and 25µg alfentanil and is administered under a 7 second period resulting in a maximal amount of 8 bolus doses per minute.

Each SVP implantation procedure is separated into four time points at which sedation scores are recorded. Patients are monitored by anaesthesia staff and SVP implantation is performed by an anaesthesiologist according to hospital protocol.

Participants are asked to fill in a written questionnaire to indicate pain score and satisfaction with the procedure when ready for discharge.

Adverse events, time consumption and operators satisfaction with implantation conditions are recorded periprocedural.

The result of this trial will provide guidance for a larger randomized trial (PACSPI-2) comparing several clinically relevant aspects of the use of PCS and local anesthesia (LA) versus LA alone during SVP implantation.

ELIGIBILITY:
Inclusion Criteria:

• Adult patients (≥18 years) scheduled for SVP implantation at Ryhov County Hospital.

Exclusion Criteria:

* Inability to operate the PCS apparatus,
* Inability to communicate in Scandinavian languages.
* Patients who require general anaesthesia or patients eligible for local anaesthesia only (i.e. severe sleep apnea).
* Propofol or alfentanil allergy.
* Intake of food (or clear fluids) within six (or two) hours prior to the procedure.
* Failure to achieve peripheral vascular access.
* Pregnancy

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients ≥18 years scheduled for SVP implantation at Ryhov County Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Participants maximal pain level | 10 minutes before discharge from recovery area
  Participants assessment of maximal pain level experienced during the procedure using a numeric rating scale from 0-10 (0=no pain, 10=worst pain I know) on patient questionnaire.

SECONDARY OUTCOMES:
Procedural time consumption | after completion of procedure
  From procedure start (local anesthesia injection) until end of procedure (last suture).
Delivered doses of propofol and alfentanil | after completion of procedure
  The total dose of given sedation and analgesia.
Grading of implantation conditions by the implanting physician | after completion of procedure
  The port-implanting physicians assessment of implantation conditions during the procedure on a numeric rating scale (0=worst possible, 10= best possible)
Participants overall satisfaction | 10 minutes before discharge from recovery area
  Participants assessment of overall satisfaction experienced during the procedure using a numeric rating scale from 0-10 (0=not satisfied at all, 10=very satisfied) on patient questionnaire
Participants satisfaction with staff | 10 minutes before discharge from recovery area
  Participants assessment of satisfaction with the staff using a numeric rating scale from 0-10 (0=not satisfied at all, 10=very satisfied) on patient questionnaire
Participants maximal pain from arm where infusion is | 10 minutes before discharge from recovery area
  Participants assessment of pain from arm with the infusion using a numeric rating scale from 0-10 (0=no pain, 10=worst pain I know) on patient questionnaire
Participants satisfaction with pain treatment during implantation | 10 minutes before discharge from recovery area
  Participants assessment of satisfaction with pain treatment on a numeric rating scale from 0-10 (0=not satisfied at all, 10=very satisfied) on patient questionnaire
Participants evaluation of the importance of receiving sedatives during the procedure | 10 minutes before discharge from recovery area
  Participants assessment of the importance of receiving sedatives on a numeric rating scale from 0-10 (0=not important, 10=very important) on patient questionnaire
Participants evaluation of the importance of being in control of sedation administration | 10 minutes before discharge from recovery area
  Participants assessment of the importance of being in control of sedation administration on a numeric rating scale from 0-10 (0=not important, 10=very important) on patient questionnaire

OTHER OUTCOMES:
Arterial puncture | after completion of procedure
  Physicians assessment after completion of procedure.
Pneumothorax | after completion of procedure
  Physicians assessment after completion of procedure.
Bradycardia | after completion of procedure
  Defined as heart < 40/minutes during the procedure
Hypoxia | after completion of procedure
  Defined as Oxygen saturation <90% or significant drop from baseline (>5% SaO2 drop) during the procedure
Airway intervention (Chin lift) | after completion of procedure
  Defined as intervention by staff with chin lift during the procedure
Respiratory rate | after completion of procedure
  Defined as respiratory rate <8/minute during the procedure
Sedation score at time points T1-T4 | during procedure at time point T1: sterile skin prepping; T2: local anaesthetic injection; T3: tunneling procedure; T4: draping removal
  Depth of sedation measured by Observer Assessment of Alertness/Sedation Scale OAAS

CONTACTS AND LOCATIONS:
Overall Officials: Margaretha Stenmarker, MD, PhD, Study Chair — Region Jönköping County
Locations (1):
- Länssjukhuset Ryhov, Jönköping, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available for sharing on request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The supporting information will be available from november 2020 until 6 months after publication
Access Criteria: Requests for sharing IPD that underlie results in a publication can be made to the principal investigator.
  The supporting information will be available on researchgate.net during the described time frame.

REFERENCES:
- [Background] Taxbro K, Hammarskjold F, Thelin B, Lewin F, Hagman H, Hanberger H, Berg S. Clinical impact of peripherally inserted central catheters vs implanted port catheters in patients with cancer: an open-label, randomised, two-centre trial. Br J Anaesth. 2019 Jun;122(6):734-741. doi: 10.1016/j.bja.2019.01.038. Epub 2019 Apr 17. PMID 31005243
- [Background] Clements W, Sneddon D, Kavnoudias H, Joseph T, Goh GS, Koukounaras J, Snow T. Randomized and controlled study comparing patient controlled and radiologist controlled intra-procedural conscious sedation, using midazolam and fentanyl, for patients undergoing insertion of a central venous line. J Med Imaging Radiat Oncol. 2018 Dec;62(6):781-788. doi: 10.1111/1754-9485.12817. Epub 2018 Oct 8. PMID 30295410
- [Background] Kreienbuhl L, Elia N, Pfeil-Beun E, Walder B, Tramer MR. Patient-Controlled Versus Clinician-Controlled Sedation With Propofol: Systematic Review and Meta-analysis With Trial Sequential Analyses. Anesth Analg. 2018 Oct;127(4):873-880. doi: 10.1213/ANE.0000000000003361. PMID 29750696
- [Background] Grossmann B, Nilsson A, Sjoberg F, Nilsson L. Patient-controlled Sedation During Flexible Bronchoscopy: A Randomized Controlled Trial. J Bronchology Interv Pulmonol. 2020 Apr;27(2):77-85. doi: 10.1097/LBR.0000000000000610. PMID 31478938
- [Result] Taxbro K, Berg S, Hammarskjold F, Hanberger H, Malmvall BE. A prospective observational study on 249 subcutaneous central vein access ports in a Swedish county hospital. Acta Oncol. 2013 Jun;52(5):893-901. doi: 10.3109/0284186X.2013.770601. Epub 2013 Feb 22. PMID 23432403
- [Derived] Seifert S, Taxbro K, Hammarskjold F. Patient-Controlled Sedation in Port Implantation (PACSPI 1) - A feasibility trial. BJA Open. 2022 Jul 31;3:100026. doi: 10.1016/j.bjao.2022.100026. eCollection 2022 Sep. PMID 37588584